CLINICAL TRIAL: NCT04484103
Title: External Validation of the Rotterdam Prostate Cancer Risk Calculator
Brief Title: RPCRC Validation Study
Acronym: PCaRisk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PCaRisk_2020
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Multivariate Risk Assessment for ISUP ≥2 Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 251 patients from the MRI-FIRST trial: The mpMRIs were performed at 16 centers with 1.5T or 3T MR units. All mpMRIs included T2-weighted imaging, diffusion-weighted imaging and dynamic contrast-enhanced imaging.
  Interventions: Other: Assessment of the diagnostic performance of the PI-RADS score (as a stand-alone) and of the RPCRC for predicting the presence of ISUP ≥2 prostate cancer at subsequent biopsy in 251 patients.

INTERVENTIONS:
Other: Assessment of the diagnostic performance of the PI-RADS score (as a stand-alone) and of the RPCRC for predicting the presence of ISUP ≥2 prostate cancer at subsequent biopsy in 251 patients. — The following features will be retrieved from the CRFs of the patients included in the MRI-FIRST trial: age, DRE findings, PSA level, prostate volume, maximal PI-RADS score; the history of biopsy will be set to a default value of "none" since all patients included in the MRI-FIRST trial were biopsy naïve.
  Then, the RPCRC will be used to calculate two different risks: the risk of "detectable prostate cancer" and of "significant prostate cancer" (ISUP ≥2) at subsequent biopsy.
  The PI-RADS score (as a stand-alone) and the risks predicted by the RPCC will be compared to the results of the prostate biopsy performed during the MRI-FIRST trial.
  Throughout the study, the version 2 of the PI-RADS score will be used.

SUMMARY:
Prostate multiparametric MRI (mpMRI) can detect ISUP ≥2 prostate cancer with high sensitivity. Adding biopsies targeting suspicious lesions seen on mpMRI to the classical 'systematic biopsies' (that sample the gland in a blinded way) improves the detection of ISUP ≥2 cancers. As a result, it is now recommended to perform a prostate mpMRI before biopsy and to combine targeted and systematic biopsy.

However, mpMRI suffers from a lack of specificity. In a recent meta-analysis, the pooled sensitivity and specificity of prostate mpMRI for detecting ISUP ≥2 cancers were 0.91 (95% confidence interval, 0.83-0.95) and 0.37 (95% confidence interval, 0.29-0.46) respectively. Thus, accurate triage of patients suitable for biopsy might not be possible using mpMRI findings alone.

The Rotterdam Prostate Cancer Risk Calculator (RPCRC) combines mpMRI results (Prostate Imaging-Reporting And Database System score) and basic clinical and biochemical data to predict the results of prostate biopsy. If validated, this tool could help selecting patients for prostate biopsy.

In this study, the investigators propose to retrospectively use the data of the prospective multicentric MRI-FIRST trial (NCT0285379) to perform an external validation of the RPCRC.

In addition, the PCaRisk study has two secondary objectives:

* To confirm that Prostate Specific Antigen density (i.e. PSA level divided by prostate volume) can stratify the risk of ISUP ≥2 cancer in patients with negative (PI-RADS 1-2) or inconclusive (PI-RADS 3) mpMRI, as suggested by recent literature
* To perform a preliminary evaluation of a lobe-specific risk calculator developed by our group and combining mpMRI results and clinical and biochemical data to predict the risk of ISUP ≥2 cancer at the lobe level.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for mpMRI and prostate biopsy due to increased PSA level, abnormal DRE or family history of prostate cancer.
* Age ≤75 years
* PSA level ≤20 ng/mL
* Clinical stage ≤T2c

Exclusion Criteria:

* Contraindication for prostate mpMRI or biopsy
* History of hip prosthesis, androgen deprivation therapy, pelvic radiotherapy or prostate cancer diagnosed after trans-urethral resection of the prostate.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the MRI-FIRST trial, i.e. biopsy-naïve patients referred for suspicion of prostate cancer on the basis of increased PSA level, abnormal DRE or family history of prostate cancer, recruited in 16 different centers in France, and who underwent mpMRI before systematic and targeted biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the Area Under Curve of the PI-RADS score and the RPCRC (significant cancer risk) for predicting ISUP ≥2 cancer at subsequent biopsy. | June 2020
  The AUC of the PI-RADS score and the RPCRC significant cancer risk will be calculated at the patient level.

SECONDARY OUTCOMES:
Comparison of the AUC of the PI-RADS score and the RPCRC (detectable cancer risk) for predicting ISUP ≥2 cancer at subsequent biopsy. | June 2020
  The AUC of the Prostate Imaging-Reporting And Data System score and the RPCRC detectable cancer risk will be calculated at the patient level.
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if PIRADS cut-off values of ≥3 and ≥4 were used as biopsy triggers | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if RPCRC detectable cancer risk cut-off values of ≥12.5% and ≥20% were used as biopsy triggers | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if RPCRC significant cancer risk cut-off value of ≥4% was used as biopsy trigger | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if biopsy was performed only in patients with a RPCRC detectable cancer risk ≥20%, or with a RPCRC detectable cancer risk ≥12.5% and a RPCRC significant cancer risk ≥4% | June 2020
AUC of PSA density in predicting ISUP ≥2 cancer at subsequent biopsy. | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if PSA density cut-off values of ≥0.15 ng/ml² and ≥0.20 ng/ml² were used as biopsy triggers | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if biopsy was performed only in patients with a PI-RADS score ≥4, or with a PI-RADS score ≤3 and a PSA density ≥0.15 ng/ml² | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and missed ISUP ≥2 cancers if biopsy was performed only in patients with a PI-RADS score ≥4, or with a PI-RADS score ≤3 and a PSA density ≥0.20 ng/ml² | June 2020
Net benefice (Decision curve analysis) for cut-off values of ≥12.5% and ≥20% for the RPCRC detectable cancer risk, of ≥4% for the RPCRC significant cancer risk, and of ≥0.15 ng/ml² and ≥0.20 ng/ml² for PSA density. | June 2020
AUC of the lobe-specific risk calculator developed by our group for predicting ISUP ≥2 cancer at subsequent biopsy. | June 2020
Number of avoided biopsies, missed ISUP 1 cancers and ISUP ≥2 cancers (at patient level) if only lobes with a lobe-specific risk of having ISUP ≥2 cancers ≥5%, ≥10% and ≥15% were biopsied. | June 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon, France